CLINICAL TRIAL: NCT05953207
Title: Evaluation of the Efficacy of Non-pharmacological Treatments for Parasomnias: a Randomized Controlled Trial
Brief Title: Non-pharmacological Treatments for Parasomnias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chantal Berna Renella (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Chantal Berna Renella, Professor, Centre de Médecine Intégrative et Complémentaire (CEMIC)
Organization: Centre de Médecine Intégrative et Complémentaire (CEMIC) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CER-VD 2023-01007
Record Dates: First submitted 2023-06-02; First posted 2023-07-20 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: NREM Parasomnia
Keywords: Medical hypnosis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical hypnosis (HYP) (Experimental): 3 medical hypnosis interventions
  Interventions: Other: Medical hypnosis
- Standard Of Care (SOC) (Active Comparator): 3 standard of care quality and sleep safety interventions
  Interventions: Other: Standard Of Care

INTERVENTIONS:
Other: Medical hypnosis — Hypnosis intervention with specific suggestions (i.e., patient's own dreamlike mentation)
  Arms: Medical hypnosis (HYP)
Other: Standard Of Care — Sleep hygiene and safety education session
  Arms: Standard Of Care (SOC)

SUMMARY:
The goal of this clinical trial is to compare the efficacy of non-pharmacological treatments (medical hypnosis and standard treatment) in patients with a non-REM parasomnia diagnosis.

Participants are randomly assigned to one of the two treatments. Treatment consists of 3 sessions. Participants receiving the standard treatment (i.e., sleep hygiene and episode risk reduction) may subsequently receive medical hypnosis.

Participation in the study involves 5 visits in total: 3 treatment visits and 2 study visits to the hospital (CHUV).

* An initial study visit to provide information and collect questionnaires prior to the start of treatment. An initial non-therapeutic hypnosis session will be carried out during electroencephalography. Estimated duration: 2h.
* A second study visit at the end of treatment, including questionnaires about your sleep and treatment. A shorter non-therapeutic hypnosis session and a second electroencephalography will be performed. Estimated duration: 1h30. This visit may also be followed by an overnight polysomnography, according to patient's choice (if performed, estimated total duration 12 hrs).

This study also involves monitoring patients' sleep for 10 nights before and after treatment: they will fill in a sleep diary and use an infrared camera.

ELIGIBILITY:
Inclusion Criteria:

* Non-REM parasomnias diagnosis according to the international classification disease of sleep disorders
* Willling and able to give informed consent
* Reporting at least one parasomniac episode per month
* Reporting at least one parasomniac episode the month prior

Exclusion Criteria:

* Refusal to use the home video recording device
* Current or planned intake (during the next 2 months) of medications/substances that may interfere with sleep architecture (e.g., hypnotics, neuroleptics, antidepressants, benzodiazepines)
* A comorbid significant somatic disease altering the brain (e.g., cancer, epilepsy, multiple sclerosis, dementia)
* A comorbid sleep disorder (e.g., apnea-hypopnea index (AHI) >= 20/hour, REM sleep behaviour disorder, restless legs syndrome with symptoms more than 2 days/week)
* A comorbid psychiatric disorder (e.g., severe depressive or anxiety disorder or psychotic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change, from pre-treatment, of mean number of parasomniac episodes at 9 weeks | Over a recording period of 10 consecutives nights, 2 weeks before (pre-treatment) and 3 weeks after (at 9 weeks) the treatment
  Parasomniac episodes scored on infrared home video recording

SECONDARY OUTCOMES:
Duration of parasomniac episodes | Over a recording period of 10 consecutives nights, 2 weeks before (pre-treatment) and 3 weeks after (at Week 9) treatment
  Using home video recording
Rate of confusional arousals, sleepwalking and sleep terrors episodes | Over a recording period of 10 consecutives nights, 2 weeks before (pre-treatment) and 3 weeks after (at Week 9) the treatment
  Categorization of parasomniac episodes' complexity (confusional arousals, sleepwalking, sleep terrors) using home video recording
Incidence of emotions related to parasomniac episodes | Through study duration, an average of 9 weeks
  Emotional impact of parasomniac episodes using questionnaires (e.g., What emotions did you feel during these episodes?; Do you have negative emotions related to your parasomnias?)
Quality of life score | At Day 0, Week 11 and Week 18
  Using a standardized questionnaire: World Health Organization Quality Of Life-BREF (WHOQOL-BREF). Score ranging from 0 to 100, higher score denoting greater perceived quality of life.
Anxiety and depression scores | At Day 0 and Week 11
  Using a standardized questionnaire: Hospital Anxiety and Depression Scale (HADS). Subscale score ranging from 3 to 21, score >8 denotes anxiety or depression.
Traumatic events score | At Day 0
  Using a standardized questionnaire: Life Event Checklist for DSM-5 (LEC-5). It does not yield a total score or a composite score.
Fatigue score | At Week 2, Week 11 and Week 18
  Using a standardized questionnaire: Pichot's fatigue scale. Score ranging from 0 to 32, score >22 denotes excessive fatigue.
Sleepiness score | At Week 2, Week 11 and Week 18
  Using a standardized questionnaire: Epworth Sleepiness Scale (ESS). Score ranging from 0 to 24, higher score denoting higher daytime sleepiness.
Sleep quality score | At Week 2, Week 11 and Week 18
  Using a standardized questionnaire: Pittsburgh Sleep Quality Index (PSQI). Score ranging from 0 to 21, higher score denoting greater acute sleep disturbances.
Severity of arousal disorders score | At Week 2, Week 11 and Week 18
  Using a standardized questionnaire: Paris Arousal Disorders Severity Scale (PADSS). Score ranging from 0 to 50, higher score denoting more severed disorders.
Circadian typology score | At Week 2, Week 11 and Week 18
  Using a standardized questionnaire: Horne & Östberg questionnaire. Score ranging from 16 to 86, higher score denoting morningness and lower score eveningness.
Changes in imagery processes | At Day 0 and Week 11
  Using power spectral sleep EEG analysis including delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), sigma (12-16 Hz), and beta (18-30 Hz) frequency bands with Titanium, Embla®, NOX-A1®.
Sleep eye movements | At Week 11 (optional)
  Using power spectral sleep EOG analysis (left and right) with Titanium, Embla®, NOX-A1®.
Sleep muscles activity | At Week 11 (optional)
  Using power spectral sleep EMG analysis (chin and anterior tibialis muscle) with Titanium, Embla®, NOX-A1®
Sleep cardiac activity | At Week 11 (optional)
  Using power spectral sleep ECG analysis (P wave, QRS complex, QT interval, PR interval...) with Titanium, Embla®, NOX-A1®.
Sleep oxygen saturation | At Week 11 (optional)
  Using sleep oxygen saturation measures with Titanium, Embla®, NOX-A1®.
Sleep airflow | At Week 11 (optional)
  Using sleep airflow measures with Titanium, Embla®, NOX-A1®.
Sleep respiratory efforts | At Week 11 (optional)
  Using abdominal and thoracic respiratory efforts measures with Titanium, Embla®, NOX-A1®.
Snoring | At Week 11 (optional)
  Using snoring measures with Titanium, Embla®, NOX-A1®.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Berna Renella, Prof, Principal Investigator — CHUV
Locations (1):
- Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland